CLINICAL TRIAL: NCT07100301
Title: Effect of a Trunk, Hip, Knee, and Ankle Exercise Program on Motor Dysfunctions Caused by Diabetic Peripheral Neuropathy: a Randomized Clinical Trial
Brief Title: Effect of an Exercise Program on Motor Dysfunctions Caused by Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, Principal Investigator, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 79226724.9.0000.0192
Record Dates: First submitted 2025-07-11; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic peripheral neuropathy; Biomechanic; Gait; Muscle strength; Kinematics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will be single-blind, so the outcome evaluator will not be aware of the allocation of participants to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal-distal group (Experimental): The experimental group will receive a proximal/distal exercise program (trunk, hip, knee and ankle).
  Interventions: Other: Proximal/distal protocol
- Distal group (Active Comparator): The control group will receive a distal exercise program (ankle and foot) available in the literature and previously tested.
  Interventions: Other: Distal protocol

INTERVENTIONS:
Other: Proximal/distal protocol — Proximal/distal exercise program (trunk, hip, knee and ankle) consisting of four stages: warm-up, strengthening, sensorimotor training and relaxation. The intervention will last 12 weeks and will take place twice a week, with an average duration of 50-60 minutes.
  Arms: Proximal-distal group
Other: Distal protocol — Distal exercise program available in the literature and previously tested. This will contain warm-up exercises, intrinsic foot muscle strengthening, extrinsic foot-ankle muscle strengthening, and functional exercises. The intervention will last 12 weeks and will take place twice a week, with an average duration of 50-60 minutes.
  Arms: Distal group

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) affects approximately half of people with Diabetes Mellitus (DM). Its repercussions on the musculoskeletal system and biomechanics mainly impact balance and locomotor function. Therefore, this study is justified by the need to design effective treatment alternatives for the motor alterations observed in people with DPN. The objective of this study will be to evaluate the effectiveness of an exercise program for the trunk, hip, knee and ankle, consisting of muscle strengthening and sensorimotor training, in the treatment of motor deficits caused by DPN. This will be a single-blind randomized clinical trial in which 64 individuals with type 2 DM and DPN will be randomly distributed between the experimental and control groups. The primary outcome will be the kinematic analysis of gait. The secondary outcomes will be: muscle strength assessed by dynamometry and the 30-second sit-to-stand test (30STS), and functional mobility through the Timed Up and Go (TUG) test. Assessments will be performed before the start of the intervention, at the end of the intervention, and at the one-month follow-up. The experimental group will perform a 12-week proximal/distal exercise program (trunk, hip, knee, and ankle). The control group will perform a distal exercise program (ankle and foot). The proposed exercise program is expected to show consistently positive results compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals aged between 45 and 75 years, male or female, diagnosed with DM2
* DPN diagnosis based on vibration sensitivity tests assessed by a 128 Hz tuning fork and tactile sensitivity measured by a 10 g monofilament
* Sedentary or irregularly active individuals (level A) according to the Physical Activity Level Classification - IPAQ
* Score of at least 5 points on the Functional Independence Measure (FIM), i.e., requires supervision, but without physical contact
* Absence of diabetic foot ulcer (DFU) for at least one month
* No amputation or at most amputation of fingers, except for the hallux

Exclusion Criteria:

* Individuals involved in physical training programs simultaneously with the intervention
* History of surgical intervention in the lower limbs or spine
* Use of walking assistance devices
* Diagnosis of severe cardiovascular disorder
* Diagnosis of other neurological impairments in addition to DPN
* Presence of dementia or inability to provide consistent information
* Severe retinopathy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  Adhesive markers will be placed at the following points on the right lower limb: greater trochanter, lateral epicondyle of the femur, lateral malleolus, and head of the fifth metatarsal. Markers will also be placed on the calcaneus of both feet. The participant will walk on a nine-meter track for filming with a digital camera. The CvMob program will be used to analyze self-selected gait speed and fast gait. Speed in m/s will be calculated based on the time it takes the participant to traverse a three-meter distance marked on the track.

SECONDARY OUTCOMES:
Joint angles during gait | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  Using adhesive markers placed on points of the right lower limb (greater trochanter, lateral epicondyle of the femur, lateral malleolus, and head of the fifth metatarsal), the angles of maximum hip flexion and extension, maximum knee flexion and extension, and maximum ankle dorsiflexion and plantar flexion will be measured from the lateral view of the right lower limb using the CvMob program.
Step length and stride | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  Using the CvMob program, stride length (cm) will be measured, which corresponds to the distance between the markers positioned on the calcaneus of the right and left feet after consecutive foot contact. Stride length will be determined by the distance in centimeters from the calcaneus marker between the first and second initial contact of the right lower limb.
Muscle strength | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  The assessment of lower limb (dominant limb) and trunk muscle strength will be performed using dynamometry. Three attempts will be performed with a minimum one-minute interval between them to avoid any fatigue effects. The highest value among the three attempts will be used as the dependent variable. The muscle groups tested will be: ankle dorsiflexors and plantar flexors, knee extensors, hip abductors, and trunk extensors.
30 second sit to stand test | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  The 30-second sit-to-stand test (30STS) is a validated test for assessing lower limb muscle strength in older adults. The patient will be asked to sit and stand in a standard-height chair (46-48 centimeters) positioned against a wall. The knees and hips should be flexed at 90 degrees, the feet flat on the floor and hip-width apart, the hands resting on the hips, and no support will be used. For 30 seconds, the participant must repeatedly sit and stand up from the chair as quickly as possible. The count will begin in the sitting position and end when the participant reaches the final standing position. The number of repetitions will be counted and recorded.

IPD SHARING:
Plan to Share IPD: No